CLINICAL TRIAL: NCT04253366
Title: A Multicentric, Single Arm, Prospective, Stratified Clinical Investigation to Evaluate the Ability of MammoWave in Breast Lesions Detection
Brief Title: Clinical Investigation to Evaluate the Ability of MammoWave in Breast Lesions Detection
Acronym: DE-17-17
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umbria Bioengineering Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DE-17-17
Record Dates: First submitted 2019-12-27; First posted 2020-02-05 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Clinical investigation with Medical Device class IIa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): All patients perform standard breast screening and also MammoWave exam.
  Interventions: Device: Clinical investigation device class IIa not marked CE

INTERVENTIONS:
Device: Clinical investigation device class IIa not marked CE — Patients should perform MammoWave exam. A short visit should be performed and during this visit a qualitative differentiation would be performed between patients with high density breast, and patients with low density breast. After the patients will be ready for the MammoWave exam. The exam will be composed of two phases: the data acquisition and the data processing. During the acquisition that should takes about 10 minutes the patients would be lying in a prone position, on a bed which is part of the MammoWave. The upper part of MammoWave has a container cup shape, which contains the breast, which also has the function of separate it from the internal parts of the device. After patient is on the bed and MammoWave would start to perform the acquisition. Once the acquisition is completed, the data will be processed through an imaging algorithm, which is integrated in the device. The final output will be composed by one or more images, plus one or more parameters describing the images.

SUMMARY:
This is a multicentric, single arm, prospective, stratified by breast density clinical investigation using Mammowave that is a device, which uses microwaves instead of ionizing radiation (X-ray)for breast lesions(BL) detection. Specifically, Mammowave employs a novel technique which generates images by processing very low power (<1 mW) microwaves. The exam takes few minutes per breast and is performed with the patient lying in a comfortable facing down position. Mammowave is safe to be used at any age, in any condition (pregnancy, specific illness) and for unlimited number of times.

DETAILED DESCRIPTION:
The number of participants will be 500 (for all the sites). The Study will be composed of two phases: a preliminary phase to 'optimize the imaging algorithm for each apparatus installed at each centre', where 15 healthy volunteers in each centre will be examined by MammoWave. In the second phase, the remaining people will be enrolled (Breast Lesions pts will be about 70% of total) and examined by MammoWave by the clinical investigator, and results will be compared with the effective diagnosis already obtained by standard clinical methods. BL includes malignant lesions (BC) and benign lesions, and may be palpable or non-palpable lesions. BL includes also isolated clustered microcalcifications.

At the end of the study, in each centre the clinical investigators will compare MammoWave output against the radiologist study output obtained using conventional exams.

In addition, at the end of the study, the MammoWave output will be centrally reviewed in blind by an independent radiologist in order to confirm the data and confirm centrally the comparisons performed locally. The primary goal of the clinical study is to assess Mammowave's ability in BL detection and differentiation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent Form
2. Women
3. Adult ≥18 years old
4. Having a radiologist study output obtained using conventional exams (such as breast specialist visit and mammography and/or ultrasound and/or magnetic resonance imaging) within the last month.
5. Patients willing to comply with study protocol and recommendations.
6. Patients with intact breast skin (i.e. without bleeding lesion, scar).

Exclusion Criteria:

1. Patients that are enrolled in another clinical study
2. Patients who belong to any vulnerable group.
3. Patients with implanted electronics.
4. Patients who have undergone biopsy less than one week before MammoWave scan
5. Patients with breast implants
6. Patients with nipple piercings (unless they are removed before MammoWave exam).
7. Participation in other studies in the last month before screening
8. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women in order to performe breast screening
Enrollment: 353 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
MammoWave sensitivity (number of 'true positive' results) | During the procedure
  MammoWave sensitivity (number of 'true positive' results) compared to Reference Standard

SECONDARY OUTCOMES:
MammoWave specificity and sensitivity (against Reference Standard) | During the baseline
  MammoWave specificity and sensitivity (against Reference Standard like Mammography, MRI and/or Echography)
Percentage of correct BL localization in terms of quadrant (against Reference Standard) | During the baseline
  Percentage of correct BL localization in terms of quadrant comparing to Reference Standard like Mammography, MRI and/or Echography
Absolute and rate agreement between different evaluator (i.e. local radiologist versus central) | Through study completion, an average of 1 year
  Absolute and rate agreement between different evaluator local radiologist versus central, in order to avoid mistakes in the MammoWave output.
Sensitivity for each breast density group | During the baseline
  Sensitivity of MammoWave according to different types of breast density groups
Sensitivity for patients which had recent mammography | During the baseline
  Sensitivity for patients which had performed recently mammography exam.
Patient satisfaction questionnaire. | During the baseline
  Patient satisfaction questionnaire output according to their experience performing MammoWave test based on 12 questions:
  n° 2 "Multiple Choice questions"
  YES, NO, explain (with open-ended text area) regarding:
  * The effective execution of MammoWave
  * The willing to promote MammoWave
    n° 5 "5 point Numeric Rating scale" ranging from 1 to 5 (1=Not at all, 5= A lot) regarding the subjective evaluation of MammoWave.
    n° 5 "3 point Numeric Rating scale" ranging from 1 to 3 (1=less, 3= more) regarding the comparative evaluation of MammoWave vs Conventional tests (Mammography, Ultrasound, Magnetic Resonance Imaging).

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Universitaria S. Martino Di Genova, Genova
- Hospital Virgen de la Salud, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No